CLINICAL TRIAL: NCT05921227
Title: Identification of Treatment Parameters the Maximize Language Treatment Efficacy for Children
Brief Title: Addressing Treatment Nonresponders
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Late Talker Phase 6; 2R01DC015642-06 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-27 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Language Development Disorders
Keywords: Late Talkers
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: All participants will start in the traditional Vocabulary Acquisition and Usage for Late Talkers (VAULT) model. Those who do not respond to treatment early on will be moved to the Augmentative and Alternative Communication Device arm of the treatment.
Who Masked: Participant, Care Provider
Masking Description: The children and their caregivers will not be told which condition they are assigned to. However, the Augmentative and Alternative Communication device is quite obvious, so although caregivers will not be explicitly told, it is likely they will be aware their child is in that arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative Treatment Including Augmentative and Alternative Communication (Experimental): Once children are shown to not respond to the usual Vocabulary Acquisition and Usage for Late Talkers (VAULT) treatment, they will be placed in this arm, which will train them to use an Augmentative and Alternative Communication device as an additional means to use to 'say' a word.
  Interventions: Behavioral: VAULT Phase 6
- Usual Vocabulary Acquisition and Usage for Late Talkers (VAULT) treatment (Active Comparator): Children who do appear to respond to treatment will continue with the full course of usual Vocabulary Acquisition and Usage for Late Talkers (VAULT) intervention.
  Interventions: Behavioral: VAULT Phase 6

INTERVENTIONS:
Behavioral: VAULT Phase 6 — VAULT is an input-based word learning intervention based on principles of statistical learning.

SUMMARY:
The goal of this clinical trial is to see if providing late talking toddlers who are not responding to the Vocabulary Acquisition and Usage for Late Talkers (VAULT) treatment with a different way of communicating will help them improve their word learning. Participants will start with VAULT word learning treatment. If, in the first few sessions, it looks like they won't respond well, they will be provided with a Big Mack Augmentative and Alternative Communication device (a button that says a word when you press it) to use for their responses. The investigators will see if this modification will help with word learning.

DETAILED DESCRIPTION:
Children will begin Vocabulary Acquisition and Usage for Late Talkers (VAULT) word learning treatment. If, after three sessions, they do not show an initial response to treatment, they will be provided with a Big Mack Augmentative and Alternative Communication device which will allow them to 'say' the treatment words with the device. Treatment will continue until the children have had 8 total weeks of treatment (2x/wk for 30 minutes per session). The investigators will measure word learning across time tracking both spoken productions and productions made with the device.

ELIGIBILITY:
Inclusion Criteria:

* Native English Speaking
* Pass pure tone hearing screening or medical report of normal hearing
* 2-3 years at start of study
* MacArthur-Bates Communicative Development Inventories (MCDI) expressive scale <10th percentile

Exclusion Criteria:

* Parental report of other diagnoses
* Enrolled in concurrent treatment elsewhere
* Nonverbal IQ <75 as measured by the Bayley Scales
* Parents unable to consistently bring child to treatment sessions.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Treatment Effect Size | Change from baseline through treatment, which will average an 8-week time frame.
  The investigators will count the number of spontaneous and probed productions of target and control words and calculate a treatment effect size (d).
Number/Rate of words learned | Change from Initial Evaluation through Follow-up, which will average a 6-month time frame.
  The investigators will measure the number of words learned and rate of words learned as reported by the parent on the MCDI starting prior to treatment and measured during, immediately following, and 4-6 weeks after the treatment.

SECONDARY OUTCOMES:
Post Treatment Retention | Change from end of treatment to follow up, which will average 4-6 weeks.
  We will use probe data or specific words and parental report to determine how many of the words the child retained from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Alt, PhD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No